CLINICAL TRIAL: NCT00318214
Title: Safety and Efficacy Study of MRE0094 to Treat Large, Single or Multiple, Chronic, Neuropathic, Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study had poor enrollment with only 16 patients randomized across 19 study centers over an 18-month period.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRE0094P-202
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Foot Ulcer, Diabetic; Diabetes Complications
Keywords: toe ulcer; heel ulcer; foot ulcer; diabetic feet; diabetic foot; complications of diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications; digital ulcers; Foot Ulcer | interventions — 2-(2-(4-chlorophenyl)ethoxy)adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MRE0094
- 2 (Placebo Comparator)
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: MRE0094 — Gel, 500 mcg/g once each day
  Arms: 1
Drug: Vehicle gel — Gel administered once per day
  Arms: 2

SUMMARY:
This is a clinical research study of an experimental topical drug for the treatment of chronic, neuropathic, diabetic foot ulcers. The purpose of the study is to determine the safety of the experimental drug when applied to large, diabetic foot ulcers. The study will also determine if the experimental drug can safely promote healing of diabetic foot ulcers better than standard treatments currently available to doctors.

Patients participating in the study may receive an active drug (MRE0094) or inactive drug (placebo). What treatment a patient will receive is determined by chance (like drawing a number from a hat). All patients will receive additional care for diabetic foot ulcers during the study.

Participation in the study can be up to 4½ months.

ELIGIBILITY:
Inclusion Criteria:

Participants included in the study must:

* Have type 1 or type 2 diabetes mellitus.
* Have problems with the nerves in their feet.
* Have a large ulcer or multiple ulcers on the bottom surface of their foot that has been present for 3 weeks or more and is of sufficient size to qualify for the study.
* Be able to apply study drug to their ulcer, or have a caregiver do it.
* Be able to visit the doctor regularly during the 4½ month study.

Exclusion Criteria:

Participants may not participate in the study if:

* Their ulcer is caused by bad blood flow to their foot.
* Their ulcer is infected.
* They cannot wear an off-loading device during the study to take pressure off the ulcer.
* They have certain other diseases, or are using certain types of drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Systemic exposure to topical MRE0094 measured by plasma concentrations of MRE0094. | Baseline (Day 1) to endpoint or 90 days, whichever is earlier
Incidence, intensity, and seriousness of adverse events (AEs). | Baseline (Day 1) to endpoint or 90 days, whichever is earlier
Changes in irritation scores. | From baseline to the various treatment visits
Changes in electrocardiograms (ECGs), vital signs, and clinical laboratory values. | Baseline, Day 50, and Day 90 (EGCs); from baseline to the various treatment visits (vital signs and lab values)

SECONDARY OUTCOMES:
Incidence of complete healing of target ulcer | At endpoint or 90 days, whichever is earlier
Time to closure and percent reduction in surface area of the target ulcer. | From baseline (Day 1) to the various treatment visits

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rolleri, Pharm.D., Study Director — King Pharmaceuticals is now a wholly owned subsidiary of Pfizer
Locations (19):
- United States (19):
  - Associated Foot & Ankle Specialists, LLC, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Roy O. Kroeker, DPM, Fresno, California
  - Innovative Medical Technologies, Los Angeles, California
  - Diabetic Foot & Wound Center, Denver, Colorado
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Karr Foot & Leg Centers, Lakeland, Florida
  - University of Miami, Miami, Florida
  - Ankle and Foot Specialist of Atlanta, Lithonia, Georgia
  - Foot Healthcare Associates, Livonia, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - North Shore Podiatry Group, Port Jefferson Station, New York
  - Calvary Hospital, The Bronx, New York
  - UNC Wound Care Clinic, Durham, North Carolina
  - Eastern Carolina Foot & Ankle Specialists, Greenville, North Carolina
  - Lehigh Valley Podiatry Associates, Allentown, Pennsylvania
  - Limb Salvage Center, Dallas, Texas
  - Southwest Regional Wound Care, Lubbock, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin